CLINICAL TRIAL: NCT00122304
Title: Safety in Hemolytic PNH Patients Treated With Eculizumab: a Multi-Center Open-Label Research Design Study
Brief Title: Study of Safety in Hemolytic Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients Treated With Eculizumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEPHERD; C04-002; NCT00133120 (obsolete NCT alias)
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Hemoglobinuria, Paroxysmal
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

INTERVENTIONS:
Drug: eculizumab

SUMMARY:
The primary objective is to evaluate the safety of eculizumab in patients with transfusion-dependent hemolytic PNH

ELIGIBILITY:
Inclusion Criteria:

* PNH > 6 months
* Type III PNH red blood cell (RBC) clone by flow cytometry >10%
* At least one transfusion in the past 2 years but no more than 3 transfusions in the past 12 months; or personal beliefs that preclude the use of transfusion with severe hemolytic PNH
* Lactate dehydrogenase (LDH) >1.5 x upper limit of normal
* Must avoid conception
* Willing and able to give written informed consent

Exclusion Criteria:

* Platelet count of <30,000/mm3
* Absolute neutrophil count <500/ul
* Active bacterial infection
* Hereditary complement deficiency
* History of bone marrow transplantation
* Participation in any other investigational drug trial or exposure to other investigational agent, device or procedure within 30 days
* Pregnant, breast-feeding, or intending to conceive
* History of meningococcal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85
Dates: Start 2004-12; Study Completion 2006-11

PRIMARY OUTCOMES:
Acceptable safety (adverse events [AEs], labs, electrocardiograms [ECGs], vital signs)
Primary surrogate of efficacy endpoint is hemolysis measured by LDH area under the curve.

SECONDARY OUTCOMES:
Hemolysis measured by the change of LDH from baseline;
Quality of Life

CONTACTS AND LOCATIONS:
Locations (48):
- United States (19):
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford University Medical Center, Division of Hematology, Stanford, California
  - Hartford Hospital, Cancer Clinical Research Office, Hartford, Connecticut
  - Cleveland Clinic Florida, Dept. of Clinical Research, Weston, Florida
  - Indiana University Cancer Pavilion, Indianapolis, Indiana
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - National Heart, Lung, and Blood Institute, National Institutes of Health, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Division of Hematology, Rochester, Minnesota
  - Washington University Medical Center, Department of Internal Medicine/Division of Hematology, St Louis, Missouri
  - Cooper University Hospital, Cooper Cancer Institute, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Division Cell Therapy, Heme Malignancies Program, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - OHSU Center for Hematologic Malignancies, Portland, Oregon
  - Presbyterian Medical Center, PENN Comprehensive Hemophilia & Thrombosis Program, Philadelphia, Pennsylvania
  - University of Utah, Hematology-BMT Department, Salt Lake City, Utah
- Australia (5):
  - Royal North Shore Hospital, Haematology Department, Saint Leonard, New South Wales
  - Princess Alexandra Hospital, Oncology Haematology Radiation Department, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Haematology/Oncology Department, Woodville South, South Australia
  - The Royal Perth Hospital, Dept. of Haematology/Level 2, Perth, Western Australia
  - Royal Melbourne Hospital, Dept. of Clinical Haematology & Medical Oncology, Parkville
- Ucl St. Luc, Hematology Department, Brussels, Belgium
- Canada (2):
  - University of Alberta, Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Centre, Clinical Research Unit Room C3080, London, Ontario
- Hopital Saint-Louis, Centre d'investigation Clinique, Paris, Cedex, France
- Germany (4):
  - Universitatsklinikum Essen, Zentrum fur Innere Medizin, Essen
  - Medizinische Hochschule Hannover, Abt. Hamatologie/Onkologie, Zentrum fur Innere Medizin, Hanover
  - Universitatskliniken des Saarlandes, Innere Medizin 1, Homburg/Saar
  - Institut fur Klinische Transfusionmedizin und Immungenetik, Abtlg. Transfusionmedizin des Univer. Ulm, Ulm
- St. James Hospital, Haematology Dept., Cancer Clinical Trial Office, Dublin, Ireland
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Dipartimento di area critica medico-chirurgica, Florence
  - Ospedale San Martino, Dept. of Hematology, Genova
  - Ospedale Maggiore di Milano, Divisione di Ematologia, Milan
  - Universita degli Studi di Napoli, Divisione di Ematologia, Azienda Universitar Policlinico, Napoli
  - Ospedale San Bortolo, Divisione di Ematologia, Vicenza
- UMC St. Radboud, Department of Hematology, Nijmegen, Netherlands
- Spain (3):
  - Hospital Clinic i Provincial, Servicio de Hematologia, Barcelona
  - Hospital Universitario Germans Trias I Pujol, Servicio de Hematologia, Barcelona
  - Hospital De La Paz, Servicio de Hematologia, Madrid
- Sweden (2):
  - Stockholm South Hospital, Division of Hematology, Stockholm
  - University Hospital, Dept. of Haematology, Uppsala
- Kantonsspital Basel, Abteilung fuer Haematologie, Basel, Switzerland
- United Kingdom (3):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Leeds General Infirmary, D Floor Brotherton Wing, Leeds
  - St. Georges Hospital, Department of Haematology, London